CLINICAL TRIAL: NCT02100306
Title: The Role of Auditory Feedback in Guiding Upper Extremity Movements
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: JCH-1234-SF
Record Dates: First submitted 2014-03-14; First posted 2014-03-31 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients (Experimental): Patients will receive:
  Auditory Feedback 100% Auditory Feedback 50% alternate
  Interventions: Behavioral: Auditory Feedback 100%; Behavioral: Auditory Feedback 50% alternate

INTERVENTIONS:
Behavioral: Auditory Feedback 100% — Patients will receive constant auditory feedback across training trials.
Behavioral: Auditory Feedback 50% alternate — Patients will receive alternating auditory feedback (1 trial auditory feedback; 1 trial no auditory feedback) across trials

SUMMARY:
Stroke is one of the leading causes of disability, with an estimated prevalence of 50,000 cases per year in Canada. Less than half of stroke patients regain use of their arm and hand. There is currently no intervention regime that is the gold standard, despite the variety of therapeutic techniques used to treat the upper extremity post-stroke. The use of external feedback to improve motor learning is a technique that has been less studied but shows promise. Therefore, the purpose of this proof of principle study it to test whether different auditory feedback frequencies can facilitate reaching ability in people with stroke. In addition brain scans will be collected that will enable us to determine how stroke severity may impact on one's ability to improve with this technique.

We hypothesize that patients who receive less feedback (50% alternate) will have enhanced learning relative to the patients who receive more feedback (100%).

ELIGIBILITY:
Inclusion Criteria:

* Unilateral first time MCA ischemic stroke
* Stroke patients should have some movement of shoulder/elbow (no movement of hand - e.g. hand, fingers - is OK)
* > 2 months post
* between 30-85 years

Exclusion Criteria:

* prior stroke
* severe comprehension (or cognitive) deficit that compromises informed consent or understanding of instructions
* contraindications to MRI (e.g. claustrophobia, metal implants)
* neurodegenerative or psychiatric disease
* apraxia
* auditory deficits that would impair testing
* prior musculoskeletal injury to back or upper extremity (including shoulder subluxation from stroke)
* skin conditions that would preclude taping of goniometers

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Change in movement error from baseline | participants will be followed for the duration of the study, an expected 3 hours per day for 2 weeks (5 days per week/10 days total)

SECONDARY OUTCOMES:
Change in range of motion | participants will be followed for the duration of the study, an expected 3 hours per day for 2 weeks (5 days per week/10 days total)
Change in movement duration | participants will be followed for the duration of the study, an expected 3 hours per day for 2 weeks (5 days per week/10 days total)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Chen, PhD, Principal Investigator — Canadian Partnership for Stroke Recovery
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- See also: Related Info — http://joycelchen.weebly.com/